CLINICAL TRIAL: NCT06545214
Title: Caracterization of the Combined Alterations in Respiration and aROUSal in Patients With Drug-resistant EpiLepsy
Acronym: CARROUSEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_1350
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; SUDEP; GTCS; Drug-resistant; Arousal; Hypercanic challenge
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Monocentric prospective non-randomized study comparing the arousal and respiratory responses to hypercapnia in adult patients with drug-resistant epilepsy and in healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with drug-resistant focal epilepsy (Other): Patients with >3 focal to bilateral tonic-clonic seizure per year and who had undergone long-term video-EEG (VEEG) monitoring for presurgical evaluation.
  After a prospective baseline, which will allow to ensure prospective seizure count for patients with epilepsy, all participants will undergo a 24-hours hospitalization. The following procedures will be carried out as part of the research:
  * Video-EEG recordings
  * Respiratory monitoring
  * Full-night polysomnography
  * 1 Hypercapnic challenge while participant is awake
  * 2 Hypercapnic challenges while participant is sleeping
  * Auditory stimulus All the medical devices used in this study are already in routine use at Hospices Civils de Lyon
  Interventions: Procedure: Video-EEG monitoring; Procedure: Respiratory monitoring and polysomnography; Procedure: 1 Hypercapnic challenge while participant is awake; Procedure: 2 Hypercapnic challenges while participant is sleeping; Procedure: Auditory stimulus; Other: Questionnaires
- Healthy subjects (Other): Selection of healthy subjects will be performed to ensure age-matching.
  After a prospective baseline, which will allow to ensure prospective seizure count for patients with epilepsy, all participants will undergo a 24-hours hospitalization. The following procedures will be carried out as part of the research:
  * Video-EEG recordings
  * Respiratory monitoring
  * Full-night polysomnography
  * 1 Hypercapnic challenge while participant is awake
  * 2 Hypercapnic challenges while participant is sleeping
  * Auditory stimulus All the medical devices used in this study are already in routine use at Hospices Civils de Lyon
  Interventions: Procedure: Video-EEG monitoring; Procedure: Respiratory monitoring and polysomnography; Procedure: 1 Hypercapnic challenge while participant is awake; Procedure: 2 Hypercapnic challenges while participant is sleeping; Procedure: Auditory stimulus; Other: Questionnaires

INTERVENTIONS:
Procedure: Video-EEG monitoring — Video-EEG monitoring
Procedure: Respiratory monitoring and polysomnography — heart rate, pulse oximetry (oxygen levels in the blood), nasal airflow, respiratory effort (thoracic and abdominal) and capnography (carbon dioxide (CO2) levels in exhaled air)
Procedure: 1 Hypercapnic challenge while participant is awake — The healthy patient/subject breathes through the mouth, using a mouthpiece and a nose clip, through a device fitted with a hermetically sealed bag that measures the various parameters of his/her breathing. At the start of the test, the healthy patient/subject breathes ambient air and his or her breathing is measured. Then, after a few minutes, the healthy patient/subject is connected to the bag, breathing in a closed circuit. This causes a gradual increase in carbon dioxide (CO2) in the inspired air. During this time, breathing parameters will be measured and gas exchanges studied with each breath. The test is stopped when the end-tidal carbon dioxide pressure (PetCO2) reaches 60 mm Hg, or in the event of intolerance.
Procedure: 2 Hypercapnic challenges while participant is sleeping — In the evening, as soon as the doctor detects on the EEG that the patient/subject is in deep sleep, various tests will be carried out to assess reactivity to wakefulness.
  Two hypercapnic challenges will be carried out during sleep, using the same procedure as for wakefulness. The test will be stopped when the healthy patient/subject wakes up, or when the end-tidal carbon dioxide pressure (PetCO2) reaches 60 mm Hg, or in case of intolerance.
Procedure: Auditory stimulus — Two auditory stimulus tests will be carried out during the patient's sleep. Using headphones, the investigator will administer auditory stimuli at regular, progressively louder intervals to determine the ability of the patient/ healthy subject to awaken to an auditory stimulus.
Other: Questionnaires — Questionnaire to assess caffeine consumption habits Quality of life questionnaires QOLIE-31 Anxiety and depression questionnaires HADS

SUMMARY:
30% of patients with epilepsy suffer from drug-resistant seizures and are at risk of epilepsy-related complications, from cognitive dysfunctions to premature mortality. Both seizures and their complications are modulated by patients' vigilance states, with a tight and bi-directional interplay between sleep and epilepsy. Several epilepsy complications are associated with sleep, such as sleep-disordered breathing or Sudden and Unexpected Death in Epilepsy (SUDEP). SUDEP is a non-traumatic death, unrelated to a documented status epilepticus, which accounts for up 50% of premature deaths in epilepsy, with a cumulative risk of ≈ 10% at 40 years in patients with childhood-onset epilepsy. SUDEP typically occurs during sleep, after a nocturnal seizure, and primarily results from a postictal central respiratory dysfunction in patients with generalized convulsive seizure (GCS), suggesting that interaction between respiratory dysfunction and sleep state may play a role in its pathophysiology.

Most of patients with drug-resistant seizures demonstrate transient peri-ictal apnea and hypoxemia, especially in the aftermath of a GCS. Experimental and clinical data suggest that most SUDEP primarily result from a fatal seizure-related respiratory arrest. In patients whose SUDEP had occurred during long-term video-EEG monitoring, we observed fatal postictal central apnea after a nocturnal GCS in all SUDEP. Accordingly, it is currently hypothesized that in a subgroup of patients, repetition of seizures may contribute to chronic alteration of respiratory regulation which may increase the risk of fatal postictal central respiratory arrest. Finally, post-mortem data in SUDEP patients showed alteration of neuronal populations involved in respiratory control in the medulla.

The complex network that regulates arousal and sleep and the respiratory network are strongly interconnected. Impairment of the interaction between central respiratory control and arousal systems has been reported in several clinical situations, including sleep apnea syndrome, sudden infant death syndrome or Prader-Willi Syndrome. In epilepsy, preclinical data in rodents indirectly support a role for 5HT in the impairment of the interactions between the arousal and respiratory systems in the cascade of events leading to SUDEP. However, no direct evidence is available, and the link between alterations of the brainstem networks involved in arousal regulation and respiratory dysfunction has not been characterized in patients with epilepsy yet.

ELIGIBILITY:
Inclusion Criteria:

Patients :

1. Written informed consent obtained from study subject and ability for study subject to comply with the requirements of the study
2. Aged 18 to 55 years old
3. Diagnosis of focal epilepsy
4. Epilepsy is refractory to treatment, as defined by the International League Against Epilepsy
5. Patients with ≥3 focal to bilateral tonic-clonic seizure (FBTCS) during the past 18 months
6. Patients who had undergone long-term video-EEG (VEEG) monitoring for presurgical evaluation in the past ten years within the Department of Functional Neurology and Epileptology at Hospices Civils de Lyon, ensuring access to detailed information about:

   * occurrence of transient respiratory dysfunction during the focal seizures, transient hypoxemia during strictly focal seizures being observed in 40% of patients(39) and in 87% of patients with at least one FBTCS during the VEEG monitoring(46)
   * localization of the epileptogenic zone, the risk of peri-ictal respiratory dysfunction being greater in seizures of temporal lobe origin than in extra-temporal seizures, even after FBTCS

Healthy subjects

1. Written informed consent obtained from study subject and ability for study subject to comply with the requirements of the study
2. Aged 18 to 55 years old

Exclusion Criteria:

Patients

1. Ongoing or chronic respiratory and/or cardiac insufficiency
2. Obstructive sleep-apnea syndrome
3. Ongoing treatment with selective serotonin reuptake inhibitor
4. Patient treated with vagal nerve stimulation
5. Pregnant women or breastfeeding women, based on declarations at V0
6. Persons receiving psychiatric care
7. Persons deprived of their liberty by a judicial or administrative decision
8. Adults subject to a legal protection measure (guardianship, curatorship)
9. Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
10. Positive urine pregnancy test at V1, if applicable

Healthy subjects

1. History of epilepsy
2. Ongoing or chronic respiratory and/or cardiac insufficiency
3. Obstructive sleep-apnea syndrome
4. Pregnant women, women in labor or breastfeeding women, based on declarations at V0
5. Persons receiving psychiatric care
6. Persons deprived of their liberty by a judicial or administrative decision
7. Adults subject to a legal protection measure (guardianship, curatorship)
8. Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
9. Positive urine pregnancy test at V1, if applicable

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
End tidal CO2 (PETCO2) value at arousal in patients with epilepsy and in healthly subjects | the night of hospitalization
  PETCO2 corresponds to the value taken at the end of a breath of the partial pressure of CO2. Two hypercapnic challenges will be performed the same night. The first will start once unequivocal N3 stage of NREM will be observed, as determined online by polysomnography data. After the termination of the first test, the patient/subject will go back to sleep and a second procedure will be performed once she/he will reach N3 stage of NREM again. Data from the two procedures will be averaged for each subject.

SECONDARY OUTCOMES:
Value of the HCVR slope during sleep in patients with epilepsy and in healthy subjects | one night of hospitalization
  HCVR measures the increase in minute ventilation (VE) induced by an increase of PETCO2. The HCVR slope, expressed in L/min/mmHg, will be calculated from the linear regression of VE and PETCO2. Data from the two procedures per night described aboves will be averaged for each subject.
  will be measured during hypercapnic sleep challenges during the night of hospitalization.
Value of the awake HCVR slope in patients with epilepsy and in healthly subjects | will be measured during hypercapnic challenges on awakening on the first day of hospitalization.
  As detailed in section 6.1.3, a hypercapnic challenge will be performed awake after arrival of the patient/subject in the epilepsy monitoring unit. Calculation of the awake HCVR slope wil be performed as described for HCVR slope during sleep
Value of the ventilatory recruitment threshold (VRT) in patients with epilepsy and in healthly subjects | will be measured during hypercapnic challenges on awakening on the first day of hospitalization.
  VRT reflects the PCO2 value at which the central chemoreflex is initiated and corresponds to the onset of compensatory and progressive rise in VE during hypercapnic challenge. The determination of VRT requires a hyperventilation baseline period during which the measured VE is the one required to maintain hypopnea under resting metabolic conditions; termed basal ventilation or the "wakefulness drive" to drive. To determine VRT, it is therefore required that the subject breathes deeply for few minutes, raising her/his tidal volume such that she/he rapidly achieves and maintaines a PETCO2 of 20-25 mmHg. Then the hypercapnic challenge can be performed. In this context, VRT can not be determined during sleep.
Number of focal to bilateral tonic-clonic seizures during the 3 months preceding the polysomnography in patients with epilepsy | Will be collected during the first day of hospitalization
Central apnea index and Obstructive Apnea Hypopnea Index | one night of hospitalization
  Sleep apneas can classified as obstructive, central or both central sleep apnea, Apnea will be defined as a decrease in peak nasal pressure of >90% of baseline, lasting at least 10 s. Hypopnea was defined as a decrease of >30% of the baseline nasal pressure, lasting at least 10 s and associated with ≥4% drop in SpO2. Central apnea will be defined by cessation > 10 seconds of airflow with simultaneous cessation of respiratory effort. The respiratory events will be scored according to the 2007 American Academy of Sleep Medicine guidelines. Apnea index will correspond to total number of each apnea type divided by total sleep time over a 24-hour period.
Sound intensity (dB) required to induced awakening | one night of hospitalization
  The paradigm will be the one proposed by Martin et al. 1996 ; Philip et al. 1994 . The stimulation will be manually delivered using earphone inserts and will consist in pure sounds of 1000Hz, from 40dB to 110dB, duration 5s. Stimulation starts after 5 min of unequivocal NREM, as assessed with continuous EEG montoring. The stimulation will start with intensity I1=50dB. If complete behavioral arousal (=awakening): stop stimulation and wait until 2 min of stable sleep (defined by re-apparition of a spindle, a K complex or REM) and next trial with I1-10dB. If arousal but no awakening: wait until 2 min of stable sleep and next trial with sound +10dB. If no Arousal : wait 10s and deliver sound +10dB or longer sound (10s)
Current and past mean daily intake of caffeine (mg/day) | Will be collected between inclusion and the first day of hospitalization
  Current usual caffeine intake and the one over the last ten years will be assessed by a validated self-survey (Simonin et al., Neuroobiology of Disease 2013) filled-in at home by the patient and, if needed, the help of the caregiver filled between the inclusion visit and the polysomnography. Its reliability, assessed by retest (mean interval: 37.5 ± 5.5 days) in 31 patients, was excellent (intraclass correlation coefficient by Fleiss method: 0.97 [95% CI: 0.94-0.98]). The mean daily intake of caffeine containing items (coffee, tea, chocolate, sodas) will be reported, along with any changes of consumption over the 10 year period. All data will be then confirmed by interview perfomed during the stay in epilepsy monitoring unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pierre Wertheimer, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No